CLINICAL TRIAL: NCT02914691
Title: Effects of Dapagliflozin Treatment on Urinary Proteomic Patterns in Patients With Type 2 Diabetes
Acronym: DapKid
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peter Rossing (Other)
Responsible Party: Sponsor-Investigator, Peter Rossing, Professor, MD, DMSc, Steno Diabetes Center Copenhagen
Organization: Steno Diabetes Center Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 2015-000335-32
Record Dates: First submitted 2016-09-09; First posted 2016-09-26 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Type 2 Diabetes; Diabetic Nephropathy
Keywords: Type 2 diabetes; Diabetic Nephropathy; Proteomics; Albuminuria; SGLT2 inhibitor
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies; Albuminuria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Active Comparator): Dapagliflozin 10 mg once daily tablet treatment
  Interventions: Drug: Dapagliflozine 10 mg once daily tablet treatment
- Placebo (Placebo Comparator): Identical once daily tablet treatment
  Interventions: Drug: Placebo identical once daily tablet treatment

INTERVENTIONS:
Drug: Dapagliflozine 10 mg once daily tablet treatment
  Arms: Active
Drug: Placebo identical once daily tablet treatment
  Arms: Placebo

SUMMARY:
Background: SGLT2 inhibitors are the first antiglycaemic drugs with a direct renal action. A part from reducing blood glucose, systemic blood pressure and albuminuria are decreased, while natriuresis is increased.

Previous research into urinary peptide patterns (proteomics) has revealed that patients in risk of progressive renal disease display a "risk peptide pattern" in their urine, ahead of decline in renal function. Furthermore a urinary proteome pattern is related to CVD risk.

The long-term impact of dapagliflozin (dapa) treatment on renal parameters is unknown, but long term randomized trials are ongoing. By investigating the impact of dapa treatment on this peptide pattern, it will be determined whether this intervention can improve the urinary proteomic peptide pattern. In addition new knowledge regarding renal processes that the treatment influences is sought.

The impact of treatment of urinary and tubular markers of oxidative stress and function (metabolomics) will be assessed. These markers are thought to represent one of several deleterious pathways involved in the pathology of diabetic renal disease, and here the impact dapa treatment will be investigated. Improvement of these markers of oxidative stress may indicate long-term benefit.

Objective: The primary objective is to assess the impact of three months of treatment with dapa 10 mg once daily or placebo on renal proteomics pattern and other risk markers of diabetic comorbidity.

Design: Double blinded, randomized, placebo-controlled crossover, single center study. Treatment period: 2 x 12 weeks.

Patient population: 40 patients with type 2 diabetes recruited from Steno Diabetes Center in accordance with the study in- and exclusion criteria.

Intervention: Dapa 10 mg daily vs. placebo. Endpoints: Primary outcome: To evaluate the effect of dapa treatment on urinary proteomic patterns in patients with type 2 diabetes, microalbuminuria and eGFR equal to or above 45 ml/min/1.73m2.

Secondary endpoints are the effect of the intervention on other markers for tubular function, inflammation, endothelial dysfunction, microcirculation, kidney function, albuminuria, vasoactive hormones in plasma, and effect on global longitudinal strain as measured by echocardiography.

Timeframe: Randomisation planned from June 2015, inclusion over the following 9 months. Last patient is expected to be completed October 2016. Data analysis completed December 2016, presentation autumn 2017 and publication early 2018.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients >18 years of age with a diagnosis of type 2 diabetes (WHO criteria).
* Patients must be on current stable antiglycaemic treatment with oral drugs (OAD) or insulin 4 weeks before start of study drug and throughout study duration.
* Patients must be on stable antihypertensive treatment (must include renin-angiotensin system blocking treatment) 4 weeks before start of study drug and throughout study duration.
* HbA1c >7.5 %
* Urinary albumin creatinine ratio (UACR) > 30 mg/g (in ≥2 out 3 morning spot urine collections prior to randomisation).
* eGFR ≥ 45 ml/min/1.73 m2
* Stable RAAS-blocking treatment (more than or equal to 4 weeks prior to visit 0) If not stable at visit 0, screening phase can be prolonged to 4 weeks.

Exclusion Criteria:

* Current treatment with loop diuretics
* Current treatment with thiazolidinediones
* Current treatment with dapagliflozin or other SGLT2 inhibitor
* Ongoing cancer treatment
* Patients on hypertension treatment who are is not on stable antihypertensive treatment (must include renin-angiotensin system blocking treatment) 4 weeks before start of study drug and throughout study duration
* Severe hepatic insufficiency and/or significant abnormal liver function defined as aspartate aminotransferase (AST) >3x upper limit of normal (ULN) and/or alanine aminotransferase (ALT) >3x ULN
* Total bilirubin >2.0 mg/dL (34.2 µmol/L)
* Positive serologic evidence of current infectious liver disease including, Hepatitis B surface antigen and antibody and Hepatitis C virus antibody
* eGFR: <45 mL/min (calculated by MDRD formula)
* History of unstable or rapidly progressing renal disease
* Volume depleted patients. Patients at risk for volume depletion due to co-existing conditions or concomitant medications, such as loop diuretics should have careful monitoring of their volume status
* Recent Cardiovascular Events in a patient:

  1. Acute Coronary Syndrome (ACS) within 2 months prior to enrolment 2.Hospitalization for unstable angina or acute myocardial infarction within 2 months prior to enrolment 3. Acute Stroke or TIA within two months prior to enrolment 4. Less than two months post coronary artery revascularization
* Congestive heart failure defined as New York Heart Association (NYHA) class IV, unstable or acute congestive heart failure. Note: eligible patients with congestive heart failure, especially those who are on diuretic therapy, should have careful monitoring of their volume status throughout the study.
* Pregnant or breastfeeding patients
* Patients who, in the judgement of the investigator, may be at risk for dehydration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-08; Primary Completion 2017-07-05 (Actual); Study Completion 2017-07-05 (Actual)

PRIMARY OUTCOMES:
Change in Urinary Peptide Patterns (Proteomics) | Up to 26 weeks
  Proteomics will be evaluated at week 0, at crossover week 12 (+/- 1 week), and at end study week 24 (+/- 1 week)

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center, Gentofte Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Larsen EL, Andersen A, Kjaer LK, Eickhoff MK, Frimodt-Moller M, Persson F, Rossing P, Lykkesfeldt J, Knop FK, Vilsboll T, Rungby J, Poulsen HE. Effects of two- and twelve-weeks sodium-glucose cotransporter 2 inhibition on DNA and RNA oxidation: two randomized, placebo-controlled trials. Free Radic Res. 2023 Feb;57(2):140-151. doi: 10.1080/10715762.2023.2213820. Epub 2023 May 19. PMID 37171199
- [Derived] Curovic VR, Eickhoff MK, Ronkko T, Frimodt-Moller M, Hansen TW, Mischak H, Rossing P, Ahluwalia TS, Persson F. Dapagliflozin Improves the Urinary Proteomic Kidney-Risk Classifier CKD273 in Type 2 Diabetes with Albuminuria: A Randomized Clinical Trial. Diabetes Care. 2022 Nov 1;45(11):2662-2668. doi: 10.2337/dc22-1157. PMID 35998283
- [Derived] Eickhoff MK, Olsen FJ, Frimodt-Moller M, Diaz LJ, Faber J, Jensen MT, Rossing P, Persson F. Effect of dapagliflozin on cardiac function in people with type 2 diabetes and albuminuria - A double blind randomized placebo-controlled crossover trial. J Diabetes Complications. 2020 Jul;34(7):107590. doi: 10.1016/j.jdiacomp.2020.107590. Epub 2020 Apr 18. PMID 32340841